CLINICAL TRIAL: NCT00408369
Title: Prophylactic Antimalarial Activity of DB289 in Volunteers Challenged With Plasmodium Falciparum
Brief Title: Prophylactic Antimalarial Activity of DB289 in Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immtech Pharmaceuticals, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C06-015
Record Dates: First submitted 2006-12-04; First posted 2006-12-06 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Prophylactic Activity Against Malaria
Keywords: prophylactic; malaria; challenge
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Drug: DB289

SUMMARY:
To evaluate the prophylactic activity of orally administered DB289 against Plasmodium falciparum in non-immune healthy volunteers who are challenged by the bite of five P. falciparum-infected Anopheles stephensi mosquitoes

DETAILED DESCRIPTION:
The primary endpoint of this study is the appearance of erythrocytic parasites (parasitemia), which indicates a prophylaxis failure. Parasitemia will be sought by multiple means, including blood culture, polymerase chain reaction (PCR), Quantitative Buffy Coat (QBC) analysis, and thick and thin blood smears (detailed methods,Appendix II).

QBC and giemsa-stained blood smears will be analyzed in real time and a positive result in any one of them is sufficient to initiate chloroquine treatment. All positive QBC analyses or blood smears will be confirmed by two experienced observers. On smears, the location of parasites will be recorded using a stage micrometer, and slides will be archived and available for later re-examination. PCR samples will be collected and stored for later analysis; cultures will be inoculated at once and maintained for 70 days.

A positive result in any one of these tests constitutes a drug failure.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* BMI between 19 and 30 (Appendix IV)
* Able to provide home address and phone number; work description, address, and phone number; and to provide the name, address, and phone number of a person willing and able to assist the investigators in making contact with the cognate volunteer during the study period
* Able and willing to follow-up intensively for 3 months of scheduled visits
* Post-menopausal or surgically sterilized women
* Score of 80% or more on a written exam to test malaria knowledge and comprehension of the study
* Serum and red cells support growth of P. falciparum in vitro (Appendix V)
* Blood type A or O
* Able and willing to provide written informed consent for screening, HIV testing, and study participation-

Exclusion Criteria:

* Clinically significant abnormalities on screening examinations

  * AST, ALT, bilirubin, hemoglobin, hematocrit, prothrombin time, partial thromboplastin time, or creatinine outside the limits of normal as defined at the time of testing by the Johns Hopkins Medical Laboratories
  * laboratory evidence of HIV infection or active viral hepatitis
  * G6PD deficiency, or hemoglobin S or C
  * Significant medical illnesses requiring systemic treatment and/or hospitalization within one month of enrollment
  * History of chronic medical illnesses, significant in the investigators' judgment
  * Self-described use of tobacco
  * History of alcohol or drug abuse
  * Use of prescribed or over-the-counter medications or nutritional supplements within two weeks of enrollment (vitamins, at or below the daily recommended dose, may be taken during the study)
  * Women of childbearing potential
  * Blood or plasma donation within 2 weeks of enrollment
  * History of malaria or residence in a malaria-endemic area
  * Allergy to mosquito bites
  * Intolerance to chloroquine, Malarone, quinine, quinidine, or tetracycline
  * Taken anti-infective drugs or quinine-containing beverages in the week prior to enrollment
  * Currently participating in other clinical trials, participated in a drug trial within two weeks of enrollment, or plan to participate in another clinical trial within three months from challenge
  * Any factors for which the investigator believes that participation of the volunteer in the study is not appropriate

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is the appearance of erythrocytic parasites
(parasitemia), which indicates a prophylaxis failure. Parasitemia will be sought by
multiple means, including blood culture, polymerase chain reaction (PCR), Quantitative
Buffy Coat (QBC) analysis, and thick and thin blood smears (detailed methods,
Appendix II).

SECONDARY OUTCOMES:
To distinguish the mechanism of prophylaxis: causal vs suppressive
To evaluate the pharmacokinetics of DB289 and DB75
To assess the safety of DB289

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A. Shapiro, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States